CLINICAL TRIAL: NCT04271553
Title: "Prepare for Operation" Bundle for Young Children Undergoing Elective Surgery: Emotional Manifestation and Anxiety
Brief Title: Home-Initiated Programme to Prepare for Operation (HIPPO) Study
Acronym: HIPPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CIRB 2017-2905
Record Dates: First submitted 2019-11-03; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Anxiety; Fear of Pain; Child Behavior
Keywords: anxiety; pre-operation
MeSH Terms: conditions — Anxiety Disorders; Child Behavior | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: prospective blinded (assessor) randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patient will undergo standard workflow for elective surgical admissions.
- Video (Experimental): In addition to standard workflow, will also receive the intervention bundle which consists of a cartoon video and sets of activity sheets
  Interventions: Other: Video

INTERVENTIONS:
Other: Video — In addition to standard workflow, participants will also receive the PFO bundle which consists of: 1) A cartoon video of about 6 minutes duration illustrating the events occurring during admission, anaesthesia and surgery and 2) Sets of activity sheets which have been tailored for different age groups. Families would be encouraged to complete activity sheets together.
  Arms: Video

SUMMARY:
A hospital admission and surgical operation commonly triggers great fear and anxiety to young children. This is caused by either lack of knowledge or misconception. Although parent and families are often given the task to prepare the child for the oncoming surgery, they often lack information and skill to accomplish this task. Although numerous measures such as pre-operative play room, parental companion during induction, distraction therapy have been employed in our institution, this remains to be a challenge for care of young surgical patients.

Our study proposes to use a "prepare-for-operation" (PFO) bundle to assist our paediatric patients and their families to prepare for surgery. The PFO bundle consists of an informative cartoon video illustrating sequence of events occurring in admission, anesthesia and surgery. The video is also accompanied by activity sheets to encourage patient and family to engage, participate and learn about all these events. They will be instructed to use this PFO bundle before admission. We believe that through this off-site and cost-effective intervention, the fear of children undergoing surgery will be significantly alleviated. The family will also have better satisfaction on hospitalization experience. If proven feasible and effective, this will be a simple intervention tool that can be made accessible to all KKH pediatric patients.

DETAILED DESCRIPTION:
Research Plan: A prospective assessor-blinded randomized controlled which will recruit 130 pediatric surgical patients aged 4-10 years, undergoing elective operation in KKH. Eligible patients will be identified when an operation date has been booked. They will be approached by a research coordinator (RC) who will counsel about the study details, and recruited after consent.

Randomisaiton will be performed. The subjects will be randomised into group A and group B.

Group A will undergo standard workflow for elective surgical admissions.

Group B, in addition to standard workflow, will also receive the PFO bundle which consists of:

A cartoon video of about 6 minutes duration illustrating the events occuring during admission, anaesthesia and surgery. Video will be given out in DVD and/or with a weblink and a QR code for scanning. The weblink is password protected and is only given to participant and their parents randomised into the video group. Instruction will be given to participants and their parents to watch the video 3 days prior to admission

Sets of activity sheets which have been tailored for different age groups. Families would be encouraged to complete activity sheets together.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 4-10 years, male or female
2. No prior surgical experience
3. Able to communicate clearly, navigate simple technical software, be awake and alert
4. Normal development
5. Able to read and communicate in English

Exclusion Criteria:

1. Abnormal development
2. Has had prior surgical experience
3. Is participating in another study

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Children's Emotional Manifestation Scale | 1 day
  the behaviour and emotional status of the child will be assessed by a blinded assessor.
  The score ranges from 5 to 25 where a score of 25 indicates 'uncooperative behaviour' and 5 indicates 'cooperative behaviour'.
Anxiety score | 1 day
  Spielberger State-Trait Anxiety Inventory Score for Children (STAIC) which is a validated anxiety score in children, or the Spielberger State-Trait Anxiety Inventory (STAI) Score which is a validated anxiety score in adolescents and adults. This score allows adjustment for the different scores that may be produced for a given situation in individuals who may vary in baseline anxiety levels.
Feeling thermometer | 1 day
  A 5-point likert scale for the child to rate their feeling, where a score of 1 indicates 'very scared' and 5 indicates 'very happy'.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | 1 day
  Presented on a 100-mm line with two extreme, "not anxious" left and "very anxious" right, on which the anesthesiologist blinded to child treatment group, marks the point that represents their perception of the child's anxiety.
Induction compliance checklist (ICC) | 1 day
  An observational scale consisting of 10 behaviors scored rated by anesthesiologist blinded to child treatment group, ranging from 0-10 where a score of 10 indicates 'very difficult child induction' and 0 indicates 'perfect/cooperative child induction'.
Admission feedback questionnaires | 1 day
  A modified version of the patient satisfaction survey currently used by KK Hospital to assess patient satisfaction with outpatient services

CONTACTS AND LOCATIONS:
Overall Officials: Li Wei Chiang, MBBS, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hosptial, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jlala HA, French JL, Foxall GL, Hardman JG, Bedforth NM. Effect of preoperative multimedia information on perioperative anxiety in patients undergoing procedures under regional anaesthesia. Br J Anaesth. 2010 Mar;104(3):369-74. doi: 10.1093/bja/aeq002. Epub 2010 Feb 1. PMID 20124283
- [Background] Burstein M, Ginsburg GS, Tein JY. Parental anxiety and child symptomatology: an examination of additive and interactive effects of parent psychopathology. [corrected]. J Abnorm Child Psychol. 2010 Oct;38(7):897-909. doi: 10.1007/s10802-010-9415-0. PMID 20432062
- [Background] He HG, Zhu L, Li HC, Wang W, Vehvilainen-Julkunen K, Chan SW. A randomized controlled trial of the effectiveness of a therapeutic play intervention on outcomes of children undergoing inpatient elective surgery: study protocol. J Adv Nurs. 2014 Feb;70(2):431-42. doi: 10.1111/jan.12234. Epub 2013 Aug 29. PMID 23991679
- [Background] Li HC. Evaluating the effectiveness of preoperative interventions: the appropriateness of using the Children's Emotional Manifestation Scale. J Clin Nurs. 2007 Oct;16(10):1919-26. doi: 10.1111/j.1365-2702.2007.01784.x. Epub 2007 Jun 30. PMID 17608635
- [Derived] Nair T, Choo CSC, Abdullah NS, Lee S, Teo LLE, Chen Y, Nah SA, Chiang LW. Home-Initiated-Programme-to-Prepare-for-Operation: evaluating the effect of an animation video on peri-operative anxiety in children: A randomised controlled trial. Eur J Anaesthesiol. 2021 Aug 1;38(8):880-887. doi: 10.1097/EJA.0000000000001385. PMID 33186309